CLINICAL TRIAL: NCT04219007
Title: Vosoritide for Selected Genetic Causes of Short Stature
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Dauber (Other)
Responsible Party: Sponsor-Investigator, Andrew Dauber, Chief of Endocrinology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013585
Record Dates: First submitted 2019-12-26; First posted 2020-01-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Short Stature
Keywords: Hypochondroplasia; SHOX Deficiency; Rasopathy; NPR2; CNP; Noonan Syndrome; Aggrecan; ACAN
MeSH Terms: conditions — Dwarfism; Hypochondroplasia; Noonan Syndrome | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Genetic Short Stature (Experimental): Vosoritide, also known as BMN 111 or modified recombinant human C-type natriuretic peptide (CNP), is a 39-amino-acid peptide analog that includes the 37 C-terminal amino acids of the human CNP53 sequence plus the addition of 2 amino acids (Pro-Gly) on the N-terminus. This structural modification conveys resistance to neutral endopeptidase (NEP) degradation, resulting in prolonged half-life (t1/2) in comparison to endogenous CNP. This increase in t1/2 allows once daily subcutaneous (SC) administration.
  Vosoritide will be administered as a single 15 μg/kg subcutaneous injection given daily for 12 months.
  Interventions: Drug: Vosoritide

INTERVENTIONS:
Drug: Vosoritide — After enrollment, subjects will be followed for a 6 month observation only period to establish a baseline height velocity as well as safety profile and quality of life assessment. Vosoritide will then be administered daily via subcutaneous injection at a dose of 15 µg/kg/day for 12 months.
  Other Names: BMN-111

SUMMARY:
Short stature can be caused by a number of genetic etiologies, many of which directly affect the growth plate. The FGFR3/CNP pathway is central to growth of the chondrocyte. The study team hypothesizes that patients with selected genetic causes of short stature that interact with this pathway will benefit from treatment with vosoritide, a CNP analog, a selective NPR-B agonist which directly targets the growth plate. This study will enroll patients with short stature in selected genetic categories and will follow them for a 6 month observation period to obtain a baseline growth velocity, safety profile and quality of life assessment. Patients will then be treated with vosoritide for 12 months and will be assessed for safety monitoring and improvement in height outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s) or guardian(s) are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure. Also, subjects under the age of 18 are willing and able to provide assent (if required) after the nature of the study has been explained and prior to performance of any research-related procedure.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age >3 years 0 days AND <10 years 364 days for males, <9 years 364 days for females
4. Pre-pubertal defined as Tanner Stage 1 breasts in females and testicular volumes <3 cc in males. This must be confirmed at the Day 1 visit prior to initiation of vosoritide.
5. Patient height <-2.25 SDS. All height SDS values are calculated using the CDC growth charts/data tables (Center for Disease Control and Prevention, 2000).
6. Patients with pathogenic or likely pathogenic variants in genes known to cause the specific genetic subgroups of short stature listed below are eligible for inclusion in the study. Pathogenicity of variants will be classified as per the American College of Medical Genetics criteria with the exception of ACAN mutations as detailed below (Richards et al., 2015). Documentation of the presence of the variant must be obtained using a lab results report from a CLIA certified laboratory. Classification of the variant's pathogenicity status will be performed by the Children's National study team.

   A. CNP deficiency due to mutations in NPPC - Subjects with heterozygous or homozygous defects in NPPC are eligible.

   B. Hypochondroplasia - Subjects with heterozygous variants in FGFR3 gene associated with hypochondroplasia are eligible. Subjects with variants in FGFR3 known to cause achondroplasia or thanatophoric dysplasia or SADDAN syndrome will be excluded. (NOTE: Hypochondroplasia cohort is closed to enrollment).

   C. Patients with heterozygous defects in NPR2 are eligible. Patients with homozygous defects in NPR2 will be excluded.

   D. Rasopathy patients (including Noonan syndrome, Costello syndrome, Cardiofaciocutaneous syndrome, Neurofibromatosis Type 1) - This include patients with heterozygous variants in the following genes:

   i. BRAF ii. CBL iii. HRAS iv. KRAS v. LZTR1 vi. MAP2K1 vii. MAP2K2 viii. MRAS ix. NF1 x. NRAS xi. PPP1CB xii. PTPN11 xiii. RAF1 xiv. RRAS xv. RIT1 xvi. SHOC2 xvii. SOS1 xviii. SOS2

   E. Patients with SHOX deficiency - Patients with either heterozygous, compound heterozygous or homozygous defects in SHOX including patients with heterozygous or homozygous deletions of the SHOX regulatory region known to cause SHOX deficiency.

   F. Patients with heterozygous defects in ACAN - Patients must be heterozygous for a mutation in the ACAN gene. As there are no validated in vitro assays that reliably assess an individual variant's effect on aggrecan function, for the purpose of this clinical trial a mutation in ACAN will be defined as:
   1. A heterozygous deletion of the entire gene or of >1 complete exons of the gene
   2. Any truncating mutation including frameshift, nonsense, splice site mutations within 2 bases of the exon/intron boundary, and start loss variants
   3. Any missense mutation which meets all of the following criteria:

   i. It has an aggregate minor allele frequency less than 1X10-5 based on the gnomAD data (gnomad.broadinstitute.org) ii. It is predicted to be damaging by BOTH Polyphen2 and SIFT iii. It segregates with the short stature phenotype in available family members or is a de novo mutation d. In-frame insertions or deletions of >1 amino acid e. In-frame insertions or deletions of 1 amino acid must meet the same criteria as missense mutations. For the prediction programs, Alanine will be substituted for the deleted amino acid.
7. Absence of growth hormone deficiency defined as an IGF-1 level above the lower limit of the normal range of the assay. The IGF-1 may be repeated during the 6 month observation period and prior to the Day 1 visit. If this repeat IGF-1 is above the lower limit of the normal range of the assay, then the subject is deemed eligible. If a patient has an IGF-1 level below the lower limit of the normal range of the assay, two growth hormone stimulation tests must be performed using the routine local protocols. Patients with a peak growth hormone level >7 ng/ml will be considered growth hormone sufficient and will be eligible for inclusion as per the Growth Hormone Research Society International consensus (Collett-Solberg et al., 2019). If indicated based on IGF-1 level from the referring clinician, the growth hormone stimulation test must be done as part of routine clinical care prior to enrollment. The rationale for using an IGF-1 below the normal range as the cut-off for further evaluation for growth hormone deficiency is that in patients with a clear genetic explanation for their short stature, an IGF-1 level anywhere within the normal range would be considered reassuring and would not lead to a growth hormone stimulation test in a routine clinical setting.
8. The subject and their guardian must speak one of the 11 languages for which the QoLISSY survey (a quality of life survey for short stature) is available. These include: English, Spanish, German, Russian, Swedish, Flemish, Italian, Turkish, French, Japanese, and Ukrainian.

Exclusion Criteria:

1. Growth plate fusion - Defined as a bone age via the Greulich and Pyle method of 13 years in females and 15 years in males. These patients have limited remaining growth potential.
2. Concomitant treatment with growth hormone or recombinant IGF-1. Patients may have been previously treated with growth hormone or IGF-1 therapy. If the patient is currently on one of these therapies, they will be required to discontinue treatment in order to begin the baseline observation period for this trial. That decision will be deferred to their treating clinical endocrinologists in conjunction with the patient's guardians. We anticipate that only patients who are having a poor response to their therapy will be interested in enrolling in the current study as there is no rationale for a patient who is receiving growth hormone therapy and having a positive response to enroll in the current study.
3. Prior treatment with a GnRH analog, aromatase inhibitor or oxandrolone
4. History of any type of malignancy
5. Chronic medical condition known to affect growth including but not limited to:

   A. Cystic fibrosis B. Diabetes C. Inflammatory Bowel Disease D. Celiac Disease E. Asthma requiring a daily inhaled steroid dose > 400 micrograms of inhaled budesonide per day or equivalent F. Taking daily oral glucocorticoids for any reason G. Note - ADHD treated with a stimulant and treated hypothyroidism with a normal TSH will NOT exclude the subject from participating in the trial.

   H. Turner Syndrome or any other chromosomal aneuploidy I. Congenital heart disease which places the subject at increased risk of an adverse cardiac outcome in the setting of hypotension including but not limited to: hypertrophic cardiomyopathy, aortic stenosis with peak gradient >50mmHg, severe aortic regurgitation (defined as pressure half time >500ms by echocardiogram), coronary insufficiency, or any anatomy with a need for an afterload reducing agent. Any patient with baseline abnormalities on echocardiogram will be reviewed with a pediatric cardiologist for appropriateness for inclusion in the study.
6. Malnutrition - Defined as a BMI <5th percentile (CDC growth charts)
7. Any clinically significant abnormality on screening tests as determined by the principal investigator. Abnormal screening labs may be repeated during the 6 month observation period prior to Day 1. If they return to normal or non-clinically significant deviations per the PI's determination, the subject may proceed with the study.
8. Known or suspected allergy to trial medication, excipients, or related products
9. The receipt of any investigational drug within 90 days prior to this trial

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events [Safety and Tolerability] | 12 months
  Number of treatment-emergent adverse events or serious adverse events per study participant
Incidence of Symptomatic Hypotension events [Safety and Tolerability] | 12 months
  Number of symptomatic hypotension events per study participant
Change from Baseline in annualized growth velocity | 12 months
  To evaluate the change from baseline in age-sex standardized annualized growth velocity in cm/year after 12 months of daily SC injections of vosoritide in patients with selected genetic causes of short stature.
Change from Baseline in standardized height SDS | 12 months
  To evaluate the change from baseline in age-sex standardized height SDS after 12 months of daily SC injections of vosoritide in patients with selected genetic causes of short stature.

SECONDARY OUTCOMES:
Changes in the seated height ratio as a measure of body proportions | 12 months
  To evaluate the seated height ratio (expressed as a percentage) as a measure of body proportions. Measurement after 12 months of treatment will be compared to baseline.
Changes in the difference between arm span and height from baseline | 12 months
  To evaluate the difference between arm span and height (measured as cm) as a measure of body proportions. Measurement after 12 months of treatment will be compared to baseline.
Changes from Baseline in bone age/chronological age | 12 months
  To evaluate changes from baseline in bone age/chronological age after 12 months of daily SC injections of vosoritide

OTHER OUTCOMES:
Characterize the area under the plasma concentration time-curve from time 0 to infinity (AUC0-∞) | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Characterize the area under the plasma concentration-time curve from 0 to the time of last measurable concentration (AUC0-t) | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Characterize maximum concentration (Cmax) of vosoritide in plasma | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Characterize the elimination half-life of vosoritide (t½) | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Characterize the apparent clearance of drug (CL/F) | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Characterize the apparent volume of distribution based upon the terminal phase (Vz/F) | 3 hours at each visit
  Estimated by non-compartmental analysis for Day 1, 6 months, and 12 months per study participant
Changes from Baseline in bone mineral density | 12 months
  To evaluate changes from baseline in bone mineral density (BMD) after 12 months of daily SC injections of vosoritide (expressed as height adjusted Z-score).
Evaluate immunogenicity and assess impact on safety and efficacy measures | 12 months
  To evaluate immunogenicity and assess impact on safety and efficacy measures after 12 months of daily SC injections of vosoritide as evidenced by rates of vosoritide antibody development, which is a standard safety metric.
Changes from baseline in quality of life after daily SC injections of vosoritide: Quality of Life of Short Stature Youth (QoLISSY) questionnaire score is expressed as a percentage | 12 months
  To evaluate changes from baseline in quality of life using the QoLISSY scale after 12 months of daily SC injections of vosoritide. The Quality of Life of Short Stature Youth (QoLISSY) questionnaire score is expressed as a percentage, with scores ranging from 0% to 100% (100% is the best score).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dauber, MS MMSc, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dauber A, Zhang A, Kanakatti Shankar R, Boucher K, McCarthy T, Shafaei N, Seaforth R, Castro MG, Dham N, Merchant N. Vosoritide treatment for children with hypochondroplasia: a phase 2 trial. EClinicalMedicine. 2024 Apr 11;71:102591. doi: 10.1016/j.eclinm.2024.102591. eCollection 2024 May. PMID 38813446